CLINICAL TRIAL: NCT05910021
Title: Early Safety and Efficiency of Interdisciplinary Laparoscopic Resection Rectopexy Combined With Sacrocolpopexy for Women With Obstructive Defecation Syndrome and Pelvic Organ Prolapse
Brief Title: Early Safety of Resection Recopy and Sacrocolpopexy
Acronym: RRPSCPcomb
Status: Completed | Type: Observational
Sponsor: Evangelisches Klinikum Köln Weyertal gGmbH (Other)
Responsible Party: Principal Investigator, Claudia Rudroff, Chief of the Department of General and visceral Surgery, Evangelisches Klinikum Köln Weyertal gGmbH
Other Study IDs: EVK KOELN; RRP_SCP_interdisciplinary (Other: EVK Köln)
Record Dates: First submitted 2023-06-10; First posted 2023-06-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Constipation by Outlet Obstruction; Pelvic Organ Prolapse; Urinary Incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with ODS and POP: This pilot study established and standardized an interdisciplinary surgical approach of laparoscopic resection rectopexy (L-RRP) combined with a laparoscopic mesh sacrocolpopexy (L-SCP) used synonymously for sacrohysteropey and sacrocervicopexy, as well. Additionally, an absorbable biological mesh (

SUMMARY:
Obstructive defecation syndrome (ODS) defines a disturbed defecation process frequently associated with pelvic organ prolapse (POP) in women. It substantially compromises quality of life and conservative treatment options are limited. In cases surgery is required the interventions are characterized by individual approaches. Laparoscopic resection rectopexy (L-RRP) combined with laparoscopic sacrocolpopexy (L-SCP) was established in an interdisciplinary setting.

DETAILED DESCRIPTION:
Obstructive defecation syndrome (ODS) defines a disturbed defecation process caused by the protrusion of the lower rectum (rectocele) or the telescoping within the rectum (intussusception). The patients must exert pressure to evacuate the rectum and manual manipulation may be required. The unsuccessful attempts to defecate are associated with a feeling of incomplete rectal voiding. ODS affects approximately 10%-25% of the population and is mainly related to female sex. The condition is frequently associated with POP. On the other hand almost 60% of the female population develop POP during their lifetime and 1/3 of them suffer bowel dysfunction. Individual aspects, such as pregnancy, childbirth, connective tissue disorders, and surgical interventions further contribute to the condition. The women experience frustration due to their disturbed defecation, compromising their quality of life substantially. Conservative treatment options are limited and do not achieve the desired long-term effect.

The surgical treatment aims at the anatomic reconstruction of the bowel and pelvic floor and has been characterized by individual approaches.

This pilot study established and standardized an interdisciplinary surgical approach of laparoscopic resection rectopexy (L-RRP) combined with a laparoscopic mesh sacrocolpopexy (L-SCP) used synonymously for all surgical reconstructions. Additionally, an absorbable biological mesh (BM) for L-SCP was offered for women who wished to preserve the uterus in cases of a planned pregnancy and those, who asked for an alternative to the synthetic mesh (SM).

* Endpoints of the study The primary study outcome parameters were the safety and efficacy of the combined laparoscopic procedure.as measured by postoperative morbidity and mortality and measured. The secondary outcome parameters were clinical and anatomical outcomes as measured by scores.
* Data management and statistical analysis The necessary clinical data were collected preoperatively, during the hospital stay, and during the follow-up examinations. All scores were documented on paper and transferred to a data bank. Data were analyzed. Quantitative variables are described as means (± standard deviation) and were compared using the Kruskal-Wallis H test and Mann-Whitney U test. Qualitative variables are summarized using count, percentage, median, and interquartile range and were compared using the Fisher's exact test. A two-sided p value of <0.05 was considered statistically significant. Because no adjustments for multiple testing were performed, the analysis were exploratory.

ELIGIBILITY:
Inclusion Criteria:

* suffering from obstructed defecation and pelvic organ prolapse
* can undergo general anesthesia
* is eligible for laparoscopic surgery

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years of age, not pregnant and suffering from the obstructed defecation disorder and a pelvic organ prolapse. Medical treatment was performed without success and surgery is needed.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Safety of the procedure | 12 months
  Complication after Surgery by Clavien Dingo Score (minimum 0=no complication, 1= complication with no intervention, 2= complication with need for medication, 3a= complication with need for intervention, 3b = need for intervention under general anesthesia, 4a = septic complication, 4b= Multiorgan failure, and maximum 5= death

SECONDARY OUTCOMES:
pelvic organ prolapse (POP) | 12 months
  POP measured by POP-Q (Score ranges from 0= no POP, 1= POP until 2 cm before the hymnal line, 2= POP reached the hymnal line, 3= POP exceeds the hymnal line, 4= full extravgtnal prolapse)
Defecation function | 12 months
  Altomare score (6 items, minimum=0, maximum = 32 points; the more points, the worse the defecation function)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Rudroff, Principal Investigator — EVK Köln Weyertal
Locations (1):
- EVK Koeln Weyertal, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request to the study coordinator.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 01.01.2024-31.12.2027
Access Criteria: Access upon request to the study coordinator.
URL: https://www.evk-koeln.de/kliniken-zentren/allgemein-und-viszeralchirurgie

REFERENCES:
- [Derived] Rudroff C, Madukkakuzhy J, Hernandez AV, Otten J, Ulrici C, Karapanos L, Ludwig S. Early safety and efficiency outcomes of a novel interdisciplinary laparoscopic resection rectopexy combined with sacrocolpopexy for women with obstructive defecation syndrome and pelvic organ prolapse: a single center study. BMC Surg. 2024 Jun 14;24(1):185. doi: 10.1186/s12893-024-02474-4. PMID 38877450